CLINICAL TRIAL: NCT00003287
Title: First Line Infusional 5-Fluorouracil, Folinic Acid and Oxaliplatin for Metastatic Colorectal Cancer or Loco-Regional Recurrency - Role of Chronomodulated Delivery Upon Survival - A Multicenter Randomized Phase III Trial
Brief Title: Combination Chemotherapy in Treating Patients With Recurrent or Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: EORTC-05963; EORTC-05963
Record Dates: First submitted 1999-11-01; First posted 2004-01-23 (Estimated); Last update posted 2012-07-02 (Estimated); Status verified 2012-06

CONDITIONS: Colorectal Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Folfox protocol; Fluorouracil; Leucovorin; Oxaliplatin

INTERVENTIONS:
Drug: FOLFOX regimen
Drug: fluorouracil
Drug: leucovorin calcium
Drug: oxaliplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. It is not yet known which regimen of combination chemotherapy is more effective in treating patients with recurrent or metastatic colorectal cancer.

PURPOSE: Randomized phase III trial to study the effectiveness of combining fluorouracil, leucovorin, and oxaliplatin in different ways in treating patients with recurrent or metastatic colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the effects of chronomodulated versus nonchronomodulated infusional administration of a 3 drug high-dose chemotherapy regimen on survival in patients with locoregionally recurrent or metastatic colorectal cancer. II. Assess the antitumor effect of the combination of fluorouracil, leucovorin calcium, and oxaliplatin given as first line chemotherapy in these patients. III. Assess the response rate and toxicity of this treatment in these patients. IV. Assess the quality of life of patients receiving this treatment.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to performance status (ECOG 0-1 vs 2), extent of liver involvement (none vs less than 25% vs 25% or greater), and institution. Patients are randomized into 2 arms: Arm I (chronotherapy): Patients receive a 4 day infusion of fluorouracil, leucovorin calcium, and oxaliplatin administered via pump using chronomodulated delivery rates. Arm II (fixed infusion rate): Patients receive leucovorin calcium and oxaliplatin as 2 hour concurrent infusions followed by fluorouracil as a 22 hour infusion on day 1. On day 2, patients receive a 2 hour infusion of leucovorin calcium followed by a 22 hour infusion of fluorouracil. For patients on both arms, courses repeat every 2 weeks until the occurrence of disease progression, severe toxicity, or complete remission for a minimum of 4 months. Quality of life is assessed prior to treatment and 2 weeks after courses 4 and 8. Patients are followed for survival.

PROJECTED ACCRUAL: A total of 554 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven locoregionally recurrent or metastatic adenocarcinoma of the colon or rectum Histologic or cytologic proof of adenocarcinoma consistent with colorectal cancer in a solitary lesion if plasma carcinoembryonic antigen level is no greater than normal Metastases not limited to bone, pleural effusion, or ascites Surgically resectable metastases not eligible No symptomatic brain metastasis At least one bidimensionally measurable lesion measuring at least 20 mm in one diameter outside a previously irradiated area

PATIENT CHARACTERISTICS: Age: 18 to 75 Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 2,000/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 3 times upper limit of normal Renal: No uncontrolled hypercalcemia Cardiovascular: No significant cardiac disease Pulmonary: No severe respiratory illness Neurologic: No peripheral sensory neuropathy Other: No uncontrolled infection or chronic disease No second malignancy except basal cell carcinoma of the skin or in situ carcinoma of the cervix

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior immunotherapy for locoregionally recurrent or metastatic colorectal cancer No concurrent prophylactic growth factor Chemotherapy: No prior chemotherapy for locoregionally recurrent or metastatic colorectal cancer At least 6 months since adjuvant chemotherapy Endocrine therapy: No prior hormone therapy for locoregionally recurrent or metastatic colorectal cancer No concurrent corticosteroids Radiotherapy: See Disease Characteristics No prior radiotherapy for locoregionally recurrent or metastatic colorectal cancer Concurrent localized analgesic radiotherapy of a bone lesion permitted unless indicative of disease progression Surgery: No prior surgery for locoregionally recurrent or metastatic colorectal cancer Other: No other concurrent investigational drug

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 554 (Estimated)
Dates: Start 1998-03; Primary Completion 2002-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francis Levi, MD, PhD, Study Chair — Institut de Cancerologie et D'Immunogenetique at Hopital Paul-Brousse
Locations (36):
- Krankenanstalt Rudolfstiftung, Vienna (Wien), Austria
- Belgium (8):
  - VZW Monica Campus Eewnfeestkliniek, Antwerp
  - Hopital Saint Jean, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels (Bruxelles)
  - Centre Hospitalier Notre Dame - Reine Fabiola, Charleroi
  - Les Cliniques Saint-Joseph ASBL, Liege (Luik)
  - CHU Sart-Tilman, Liège
  - Clinique Sainte Elisabeth, Namur
  - Centre Hospitalier de Lorraine, Virton
- Canada (2):
  - Sunnybrook and Women's College Health Sciences Centre, North York, Ontario
  - Centre Hospitalier Regional de Rimouski, Rimouski, Quebec
- France (14):
  - Centre Hospitalier de la Cote Basque, Bayonne
  - Centre Jean Perrin, Clermont-Ferrand
  - Clinique du Parc, Croix
  - Centre de Lute Contre le Cancer,Georges-Francois Leclerc, Dijon
  - Hopital Perpetuel Secours, Levallois-Perret
  - Centre Oscar Lambret, Lille
  - Centre Hospital Regional Universitaire de Limoges, Limoges
  - Hopital Notre-Dame de Bon Secours, Metz
  - Centre Hospitalier de Montlucon, Montluçon
  - Clinique Hartmann, Neuilly-sur-Seine
  - Hopital Cochin, Paris
  - Centre Rene Huguenin, Saint-Cloud
  - Hopital Bellevue, Saint-Etienne
  - Hopital Paul Brousse, Villejuif
- Klinikum der Friedrich-Schiller Universitaet Jena, Jena, Germany
- University Hospital of Heraklion, Iraklion (Heraklion), Crete, Greece
- Italy (6):
  - Universita G.D'Annunzio Di Chieti, Chieti
  - Azienda Ospedale S. Luigi - Universita Di Torino, Orbassano, (Torino)
  - Fondazione Salvatore Maugeri, Pavia
  - Azienda Ospedaliera "Santa Maria Degli Angeli", Pordenone
  - Ospedale Oncologico Regionale, Rionero in Vulture
  - Istituti Fisioterapici Ospitalieri - Roma, Rome
- Haukeland Hospital - University of Bergen, Bergen, Norway
- Portugal (2):
  - Hospital Fernando Fonseca, Amadora
  - Hospital De Santo Antonio Dos Capuchos, Lisbon (Lisboa)

REFERENCES:
- [Background] Efficace F, Innominato PF, Bjarnason G, Coens C, Humblet Y, Tumolo S, Genet D, Tampellini M, Bottomley A, Garufi C, Focan C, Giacchetti S, Levi F; Chronotherapy Group of the European Organisation for Research and Treatment of Cancer. Validation of patient's self-reported social functioning as an independent prognostic factor for survival in metastatic colorectal cancer patients: results of an international study by the Chronotherapy Group of the European Organisation for Research and Treatment of Cancer. J Clin Oncol. 2008 Apr 20;26(12):2020-6. doi: 10.1200/JCO.2007.12.3117. PMID 18421055
- [Background] Giacchetti S, Zidani R, Perpoint B, et al.: Phase III trial of 5-fluorouracil (5-FU), folinic acid (FA), with or without oxaliplatin (OXA) in previously untreated patients (pts) with metastatic colorectal cancer (MCC). [Abstract] Proceedings of the American Society of Clinical Oncology 16: A805, 229a, 1997.
- [Background] Levi F, Zidani R, Misset JL. Randomised multicentre trial of chronotherapy with oxaliplatin, fluorouracil, and folinic acid in metastatic colorectal cancer. International Organization for Cancer Chronotherapy. Lancet. 1997 Sep 6;350(9079):681-6. doi: 10.1016/s0140-6736(97)03358-8. PMID 9291901
- [Background] Mormont MC, Bleuzen P, Lellouch J, et al.: Prognostic value of circadian rhythm assessment for survival of patients with metastatic colorectal cancer. [Abstract] Proceedings of the American Society of Clinical Oncology 16: A-956, 269a, 1997.
- [Result] Innominato PF, Giacchetti S, Moreau T, Smaaland R, Focan C, Bjarnason GA, Garufi C, Iacobelli S, Tampellini M, Tumolo S, Carvalho C, Karaboue A, Levi F; ARTBC International Chronotherapy Group. Prediction of survival by neutropenia according to delivery schedule of oxaliplatin-5-Fluorouracil-leucovorin for metastatic colorectal cancer in a randomized international trial (EORTC 05963). Chronobiol Int. 2011 Aug;28(7):586-600. doi: 10.3109/07420528.2011.597532. PMID 21859417
- [Result] Giacchetti S, Bjarnason G, Garufi C, Genet D, Iacobelli S, Tampellini M, Smaaland R, Focan C, Coudert B, Humblet Y, Canon JL, Adenis A, Lo Re G, Carvalho C, Schueller J, Anciaux N, Lentz MA, Baron B, Gorlia T, Levi F; European Organisation for Research and Treatment of Cancer Chronotherapy Group. Phase III trial comparing 4-day chronomodulated therapy versus 2-day conventional delivery of fluorouracil, leucovorin, and oxaliplatin as first-line chemotherapy of metastatic colorectal cancer: the European Organisation for Research and Treatment of Cancer Chronotherapy Group. J Clin Oncol. 2006 Aug 1;24(22):3562-9. doi: 10.1200/JCO.2006.06.1440. PMID 16877722
- [Result] Garufi C, Bjarnason GA, Giacchetti S, et al.: Independent prognostic value of the rest/activity circadian rhythm on overall survival (OS) in patients (pts) with metastatic colorectal cancer (MCC) receiving first line chemotherapy with 5-fluorouracil, leucovorin and oxaliplatin: a companion study to EORTC 05963. [Abstract] J Clin Oncol 23 (Suppl 16): A-3553, 259s, 2005.
- [Result] Innominato PF, Focan C, Bjarnason GA, et al.: Quality of life (QoL) correlates with the rest/activity circadian rhythm (RAR) in patients (pts) with metastatic colorectal cancer (MCC) on first line chemotherapy with 5-fluorouracil, leucovorin and oxaliplatin : an international multicenter study (EORTC 05963). [Abstract] J Clin Oncol 23 (Suppl 16): A-8029, 736s, 2005.
- [Result] Lévi F, Gorlia T, Tubiana N, et al.: Gender as a predictor for optimal dynamic scheduling of oxaliplatin, 5-fluorouracil and leucovorin in patients with metastatic colorectal cancer. Results from EORTC randomized phase III trial 05963. [Abstract] J Clin Oncol 23 (Suppl 16): A-3587, 267s, 2005.
- [Result] Giacchetti S, Bjarnason GA, Garufi C, et al.: First line infusion of 5-fluorouracil, leucovorin, oxaliplatin for metastatic colorectal cancer chronomodulated versus conventional delivery. A multicenter randomized trial of the EORTC chronotherapy group. [Abstract] Proceedings of the American Society of Clinical Oncology 21: A-2231, 2002.